CLINICAL TRIAL: NCT05233943
Title: Investigation of the Effects of Trunk Position Sense and Spinal Posture on Balance Function in Parkinson's Patients
Brief Title: The Relationship of Trunk Position Sense and Spinal Posture With Balance in Parkinson's
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Ertuğrul Yaşa, Assoc. Prof, Gulhane School of Medicine
Other Study IDs: 2022-48
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; Postural Kyphosis, Lumbosacral Region; Postural Kyphosis; Postural Lordosis, Lumbosacral Region; Balance; Distorted
Keywords: Proprioception; Parkinson Disease; Posture
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's patients: The cognitive function of Parkinson's patients will be assessed using the "Standardized Mini Mental Test " .
  The spinal posture will be evaluated using "IDIAG M360 Spinal Mouse " .
  Parkinson's patients' spinal position sense will be assessed using a "repositioning error test" with J-TECH medical, Salt Lake City, USA Dual Digital Inclinometer.
  Dynamic and static components of the balance function will be evaluated with 'four square step tests' and 'stand on one leg' tests respectively
  Interventions: Device: Spinal Mouse and Digital Inclinometer
- Healthy control group: The cognitive function of Parkinson's patients will be assessed using the "Standardized Mini Mental Test " .
  The spinal posture will be evaluated using "IDIAG M360 Spinal Mouse " .
  Parkinson's patients' spinal position sense will be assessed using a "repositioning error test" with J-TECH medical, Salt Lake City, USA Dual Digital Inclinometer.
  Dynamic and static components of the balance function will be evaluated with 'four square step tests' and 'stand on one leg' tests respectively
  Interventions: Device: Spinal Mouse and Digital Inclinometer

INTERVENTIONS:
Device: Spinal Mouse and Digital Inclinometer — The spinal mouse device is non-invasive and does not have any danger. The posture is evaluated by moving from top to bottom on the spine of the person. Data on the device is transferred to the computer via Bluetooth. The person's posture is evaluated in the sagittal plane by making maximum flexion, neutral stance and maximum extension positions, and in the frontal plane by lateral flexion to the right and left.
  Digital Inclinometer; It is a non-invasive measurement tool that investigators measure the position sense of the body, which has two parts, one fixed and one movable. The immobile part of the digital inclinometer is placed at the sacrum and the movable part is placed at the T4 spine level. The person is made 30 degrees of trunk flexion. Then, he is expected to perform 5 repetitions of 30 degrees of trunk flexion with his eyes closed. Deviation angles are recorded.
  Other Names: Four Square Step Tests; One Leg Stance Test

SUMMARY:
The 4 main motor symptoms seen in Parkinson's patients are tremor, rigidity, postural instability and bradykinesia. In addition to these, another common symptom investigators encounter is balance problems. Increasing balance problems can lead to falls and fractures over time, which will further reduce the independence of Parkinson's patients who are not already active enough and reduce their quality of life. For these reasons, it is very important that balance is achieved and sustainable. It has been found in previous studies that spinal posture and body position sensation are affected in Parkinson's patients. But to our knowledge, no study has been found in the literature to address the effect these have had on balance function. In our planned study, investigators aim to investigate the effects of spinal posture and body position sensation on balance function.

DETAILED DESCRIPTION:
Resting tremor, muscular rigidity, bradykinesia (slowing of movements) and postural instability in Parkinson's patients constitute the 4 main motor symptoms of Parkinson's. In addition, he has been in various studies where posture is affected in Parkinson's disease and proprioceptive sensory loss is seen. These symptoms reduce the quality of life of patients and can also cause loss of balance. It is very important to maintain balance due to problems such as loss of balance in Parkinson's patients leading to falls and the resulting fractures. Determining the factors that may cause falls in Parkinson's patients is important because of its guidance in terms of preventive approaches and treatment options to be developed afterwards. In our research in literature, no study has been found in Parkinson's exploring the effects of spinal proprioceptive sensory loss and spinal posture on balance function. With this work planned accordingly:

(A) Loss of spinal proprioceptive sensation in Parkinson's, (B) Changes in spinal posture in Parkinson's and (C) It was intended to investigate the effects of spinal proprioceptive sensory loss and spinal postural changes on balance function in Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria For Parkinson's patients:

* Being 18 years or older
* Receiving a diagnosis of Parkinson Disease made by a specialist neurologist
* Being able to walk independently
* Being between stages 1-4 on the Hoehn & Yahr scale

Inclusion Criteria For Healthy Volunteers :

-Being 18 years or older

Exclusion Criteria For Parkinson's patients:

* Having any neurological disease other than Parkinson's
* Presence of cardiovascular, vestibular and musculoskeletal disease
* Having a score of <24 on the Standardized Mini Mental Test

Exclusion Criteria For Healthy Volunteers :

* Having any disease that may affect balance, gait, posture and respiratory functions
* Using sedative - antidepressant medication that will impair physical well-being
* Having a score of <24 on the Standardized Mini Mental Test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals with similar age and body mass index values for Parkinson's patients who were diagnosed with Parkinson's disease according to the UK Parkinson's Disease Association Brain Bank criteria, followed in the Health Sciences University Gülhane Training and Research Hospital Neurology Department Parkinson's Polyclinic, and the control group will be included in the study. After the participants are informed about the study, a signed informed consent form will be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Balance function | 30.02.2022
  The balance function of the person is evaluated with the four-square step test and the one-leg stance tests. In the test with 4 squares, the person takes a step forward, sideways and backwards, both clockwise and counterclockwise, by coming into the square. While the person is on his right foot, he raises his left foot and is asked to stand on one foot as long as he can stand. Then the reverse is done. The times of these two tests are recorded with a stopwatch.

SECONDARY OUTCOMES:
Spinal Posture | 30.03.2022
  Spinal posture in the sagittal and frontal planes of the spine is evaluated for kyphosis, lordosis, and scoliosis.
Trunk Position Sense | 30.03.2022
  With the repositioning error test, the trunk is flexed to 30 degrees and the deviation angles of the person are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No